CLINICAL TRIAL: NCT02995551
Title: Danish Rct on Exercise Versus Arthroscopic Meniscal Surgery for Young Adults (DREAM) - A Randomized Controlled Trial of Meniscal Tear Treatment in Young Adults
Brief Title: Danish Rct on Exercise Versus Arthroscopic Meniscal Surgery for Young Adults
Acronym: DREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Copenhagen University Hospital, Hvidovre (Other); Aalborg University Hospital (Other); Sygehus Lillebaelt (Other); Naestved Hospital (Other); Odense University Hospital (Other); Slagelse Hospital (Other); Danish Council for Independent Research (Other); IMK Almene Fond (Other); Lundbeck Foundation (Other); The Danish Rheumatism Association (Other); Spar Nord Foundation (Unknown); Association of Danish Physiotherapists (Other); Regionshospitalet Silkeborg (Other)
Responsible Party: Principal Investigator, Søren Thorgaard Skou, PT, PhD, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20160151; DFF - 6110-00045 (Other Grant/Funding Number: Danish Council for Independent Research)
Record Dates: First submitted 2016-12-08; First posted 2016-12-16 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Tear of Meniscus of Knee
Keywords: Menisci, Tibial; Knee Injuries; Arthroscopy; Exercise; Young adults; Treatment Outcome; Humans
MeSH Terms: conditions — Knee Injuries; Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthroscopy (Experimental): Arthroscopic meniscal repair or resection will be conducted at the discretion of the operating surgeon (this cannot be determined before the surgeon has visual confirmation about the exact knee pathology and extend of the meniscal tear by scope).
  Interventions: Procedure: Arthroscopic meniscal repair or resection
- Exercise and Education (Active Comparator): Patients allocated to exercise therapy and education will participate in a 12-week (2 exercise sessions per week) supervised neuromuscular and strengthening exercise program tailored to 18-40 years old patients with a meniscal tear. Furthermore, they will participate in a patient education program developed through interviews with pilot study participants, from our experiences from the Good Life with osteoArthritis in Denmark (GLA:D) program for patients with knee and hip pain. Both the exercise and education will take place in a number of private physiotherapy clinics associated with the GLA:D program, specifically trained to supervise and lead the treatment in this study.
  Interventions: Behavioral: Exercise and education

INTERVENTIONS:
Procedure: Arthroscopic meniscal repair or resection — Arthroscopic meniscal repair or resection following standard procedures.
  Arms: Arthroscopy
Behavioral: Exercise and education — A 12-week (2 exercise sessions per week) supervised neuromuscular and strengthening exercise program tailored to 18-40 years old patients with a meniscal tear combined with patient education teaching the participants about their disease and how to manage it through exercise and in their daily life.
  Arms: Exercise and Education

SUMMARY:
There are two cartilage structures in each knee joint called a meniscus. A torn meniscus can be caused by either a smaller or larger trauma or be a degenerative age-related tear. Arthroscopic meniscal surgery is the most common orthopedic procedure, but no high-quality studies have investigated the efficacy of meniscal surgery for younger patients (i.e. 40 years or younger) in comparison to non-surgical treatments.

The purpose of this study is to determine if a strategy of early arthroscopic meniscal surgery (repair or resection) is superior to a strategy of initial individualized supervised exercise therapy including patient education with the option of later surgery if needed in improving pain, function and quality of life in young patients (18-40 years) with meniscal tears.

The hypothesis is that patients treated with early arthroscopic meniscal surgery will improve more than patients treated with exercise and education.

DETAILED DESCRIPTION:
Arthroscopic meniscal surgery is the most common orthopedic procedure. In Denmark, meniscal surgeries have doubled from around 9.000 yearly procedures in 2000 to more than 17.000 in 2011, with the total number of meniscal surgeries exceeding 150.000 in this period. Similar trends have been observed in the US, where more than 700.000 orthopedic procedures are carried out annually. Numerous randomized controlled trials (RCT) have investigated the efficacy of meniscal surgery compared with placebo surgery, in addition to non-surgical treatment and in direct comparison to exercise in middle-aged and older patients.

However, no RCTs have investigated the efficacy of meniscal surgery for younger patients (i.e. 40 years or younger) in comparison to non-surgical treatments. In contrast to middle-aged and older adults with degenerative meniscal tears of unknown origin, most tears in younger adults (18-40 years) are of traumatic origin (i.e. such as a sports related trauma), which highlights the need for a high-quality trial in the younger population.

The aim of this RCT is to investigate if early arthroscopic meniscal surgery (repair or resection) is superior to individualized supervised exercise therapy and education, with the option of later surgery if needed, in improving pain, function and quality of life in young patients (18-40 years) with meniscal tears. The study hypothesis is that patients randomized to surgery will improve significantly more in pain, function and quality of life after 12 months than those randomized to exercise and education.

Patients fulfilling eligibility criteria and willing to participate in the study will be randomized to one of the two groups after the baseline assessment with follow-up after 3, 6 and 12 months (Subsequently, a 24-month follow-up has been added):

1. Arthroscopic meniscal surgery: Arthroscopic meniscal repair or resection will be conducted at the discretion of the operating surgeon (this cannot be determined before the surgeon has visual confirmation about the exact knee pathology and extend of the meniscal tear by scope).

   After surgery, patients will receive the standard rehabilitation in the postoperative period depending of type of surgery, since this differs for patients who have had resection and repair. A standard folder with exercises will be given to those having a partial meniscectomy to ensure a minimum level of rehabilitation after the surgery across the hospitals.
2. Exercise therapy and patient education: Patients allocated to exercise therapy and education will participate in a 12-week (2 exercise sessions per week) supervised neuromuscular and strengthening exercise program tailored to 18-40 years old patients with a meniscal tear. Furthermore, they will participate in a patient education program developed through interviews with pilot study participants, from our experiences from the Good Life with osteoArthritis in Denmark (GLA:D) program for patients with knee and hip pain. Both the exercise and education will take place in a number of private physiotherapy clinics associated with the GLA:D program, specifically trained to supervise and lead the treatment in this study. A similar exercise program and educational program have been shown to be effective in improving pain, function and quality of life in patients with other types of knee injuries and knee pain.

Observational cohort:

Patients fulfilling all eligibility but unwilling to participate in the randomized study and patients 18-40 years of age with a clinical history and symptoms consistent with a meniscal tear that does not fulfill the other criteria are asked to participate in an observational cohort with the same questionnaires as in the RCT, but following usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 40 years with knee pain
* Clinical history and symptoms consistent with meniscal tear and meniscal tear verified on magnetic resonance imaging (MRI)
* Deemed eligible for meniscal surgery (i.e. repair or resection) by the examining orthopedic surgeon
* Willing to participate in 12 weeks of supervised exercise twice a week or undergo surgery for the meniscal tear as soon as possible

Exclusion Criteria:

* Previous knee surgery on the affected knee
* Clinical suspicion (acute locking of knee AND/OR extension deficit) of displaced bucket-handle tear confirmed by MRI
* Fracture of the affected extremity within the previous 12 months
* Complete rupture of one or more knee ligaments.
* Participation in supervised systematic exercise for knee problems within the last 3 months prior to recruitment
* Other reasons for exclusion (Unable to understand Danish, mentally unable to participate, etc.)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
the Knee Injury and Osteoarthritis Outcome Score (KOOS4) | Primary endpoint: Change from baseline to 12 months.
  The mean score for the KOOS subscales Pain, Symptoms, Function in sports and recreational activities, and Quality of life. All visits (baseline, 3, 6 and 12 months) will be included in the analysis. Will also be assessed after 24 months.

SECONDARY OUTCOMES:
The five KOOS subscales | Primary endpoint: Change from baseline to 12 months.
  To allow for clinical in-depth interpretation, the primary outcome will be complemented by subscale scores from each of the five individual KOOS subscales. All visits (baseline, 3, 6 and 12 months) will be included in the analysis. Will also be assessed after 24 months.
Western Ontario Meniscal Evaluation Tool (WOMET) | Primary endpoint: Change from baseline to 12 months.
  WOMET is a meniscus specific patient-reported outcome measure that will be used to complement the KOOS score. All visits (baseline, 3, 6 and 12 months) will be included in the analysis. Will also be assessed after 24 months.
Isometric muscle strength | Primary endpoint: Change from baseline to 3 months.
  Isometric muscle strength will be assessed using the FysioMeter. Assessed at baseline, 3 and 12 months.
The maximum number of knee-bends in 30s | Primary endpoint: Change from baseline to 12 months.
  The maximum number of knee-bends in 30s is one of three measures of functional performance. All visits (baseline, 3, 6 and 12 months) will be included in the analysis.
The one-leg hop for distance | Primary endpoint: 12 months.
  The one-leg hop for distance is one of three measures of functional performance. Assessed only at 12 months.
The 6 m timed hop | Primary endpoint: 12 months.
  The 6 m timed hop is one of three measures of functional performance. Assessed only at 12 months.
Adverse events | Primary endpoint: 12 months.
  Adverse events (AE) and serious adverse events (SAE) will be recorded at all follow-ups by asking the participants about potential AEs using open-probe questioning to ensure that all AEs are recorded. Furthermore, the medical records from the participating hospitals will be checked at the primary endpoint (12 months) for all AEs occurring from inclusion until the 12 months follow-up. AEs will be categorized into index knee or other sites and will be recorded and assessed for severity independent of whether or not there is a causal relationship with study treatments. Assessed at 3, 6 and 12 months. Will also be assessed after 24 months.
Structural knee joint changes | Baseline to 24 months
  Structural knee joint changes from baseline to 24 months will be assessed using the Anterior Cruciate Ligament OsteoArthritis Score (ACLOAS).

OTHER OUTCOMES:
EQ-5D | Primary endpoint: Change from baseline to 12 months.
  General health will be assessed using the EQ-5D-5L questionnaire (5-level version), both the descriptive index and the EQ-VAS. This will also allow for a later cost-effectiveness analysis. Assessed at baseline, 3, 6 and 12 months. Will also be assessed after 24 months.
Questions on function with Short Message Service (SMS) | Each week during the first 3 months and after that each month until the 12 months follow-up
  The subscale Sport/Rec from the KOOS
Questions on pain with Short Message Service (SMS) | Each week during the first 3 months and after that each month until the 12 months follow-up
  Pain intensity going up/down stairs and pain intensity during sitting/lying on a 11-point Numeric Rating Scale (NRS)
Physical activity level | Primary endpoint: 12 months. Assessed at baseline, 3, 6 and 12 months. Will also be assessed after 24 months.
Participation in sports (Tegner activity scale) | Primary endpoint: 12 months. Assessed at baseline, 3, 6 and 12 months. Will also be assessed after 24 months.
Global Perceived Effect (GPE) | Primary endpoint: 12 months.
  Answered on 7-point Likert scale. Assessed at 3, 6 and 12 months. Will also be assessed after 24 months.
Patient Acceptable Symptom State (PASS) | Primary endpoint: 12 months.
  "When you think of your knee function, will you consider your current condition as satisfying? By knee function, you should take into account your activities of daily living, sport and recreational activities, your pain and other symptoms and your quality of life". Answered by "yes" or "no". Assessed at 3, 6 and 12 months. Will also be assessed after 24 months.
Patient-reported treatment failure. | Primary endpoint: 12 months. Will also be assessed after 24 months.
  Only answered by patients answering "no" to PASS. "Would you consider your current state as being so unsatisfactory that you consider the treatment to have failed?". Answered by "yes" or "no".
Patient-reported mechanical symptoms related to the knee | Assessed at baseline, 3, 6 and 12 months.
  Patient-reported mechanical symptoms, i.e. catching and locking of the knee. Presence and frequency answered on 5-point scale.
Knee instability | Assessed at baseline, 3, 6 and 12 months. Will also be assessed after 24 months.
  Patient-reported knee instability. Presence and frequency of knee instability answered on a 6-point scale and how much it affects activity level answered on a 6-point scale.
Compliance with exercise (only for patients in the exercise group) | Assessed at 3 months
  The number of exercise sessions that the patient participate in out of the total 24 supervised sessions.
Patient-reported participation in post-surgery exercise (only for patients in the surgery group) | Assessed at 3 months
  Supervised or unsupervised and number of sessions.
Surgery and other treatments during follow-up | Primary endpoint: 12 months.
  Assessed at baseline, 3, 6 and 12 months by self-report and review of medical journals (surgery only). Other knee surgery will also be assessed at 24 months.
Pain intensity on a 11-point Numeric Rating Scale (NRS) | Assessed at 3 months
  Before and after each of the 24 supervised exercise sessions the patients will report their pain intensity. Only the patients in the group randomized to exercise and education.
Expanded version of the International Society of Arthroscopy, Knee Surgery and Orthopedic Sports Medicine (ISAKOS) classification of meniscal tears questionnaire | Day 1 after surgery
  Information about location of tear, type of tear and type of treatment (repair or resection) will be collected using an expanded version of the International Society of Arthroscopy, Knee Surgery and Orthopedic Sports Medicine (ISAKOS) classification of meniscal tears questionnaire by the operating surgeon. This will be supplemented with data from surgery reports.

CONTACTS AND LOCATIONS:
Overall Officials: Søren T. Skou, PT, PhD, Principal Investigator — University of Southern Denmark and Næstved-Slagelse-Ringsted Hospitals; Jonas B Thorlund, MSc, PhD, Study Chair — University of Southern Denmark; Martin Lind, Prof, MD, PhD, DMSc, Study Chair — Aarhus University Hospital; Per Hölmich, Prof, MD, DMSc, Study Chair — Copenhagen University Hospital, Amager-Hvidovre; Hans P Jensen, MD, Study Chair — Aalborg University Hospital; Carsten Jensen, MSc, PhD, Study Chair — Lillebælt Hospital in Kolding; Muhammad Afzal, MD, Study Chair — Naestved Hospital; Uffe Jørgensen, Prof, MD, DMSc, Study Chair — Odense University Hospital; Mogens Strange Hansen, MD, PhD, Study Chair — Elective Surgery Centre, Regionshospitalet Silkeborg
Locations (7):
- Denmark (7):
  - Department of Orthopedic Surgery, Aalborg University Hospital, Aalborg
  - Department of Sports Traumatology, Aarhus University Hospital, Aarhus
  - Department of Orthopedic Surgery, Copenhagen University Hospital, Amager-Hvidovre, Copenhagen
  - Department of Orthopedic Surgery, Lillebælt Hospital in Kolding, Kolding
  - Department of Orthopedic Surgery, Næstved Hospital, Næstved
  - Department of Orthopedics and Traumatology, Odense University Hospital, Odense
  - Elective Surgery Centre, Regionshospitalet Silkeborg, Silkeborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skou ST, Holmich P, Lind M, Jensen HP, Jensen C, Garval M, Thorlund JB. Early Surgery or Exercise and Education for Meniscal Tears in Young Adults. NEJM Evid. 2022 Feb;1(2):EVIDoa2100038. doi: 10.1056/EVIDoa2100038. Epub 2022 Jan 25. PMID 38319181
- [Derived] Clausen SH, Skou ST, Boesen MP, Radev DI, Kurt EY, Damsted C, Holmich P, Lind M, Torring S, Isaksen C, Varnum C, Englund M, Thorlund JB. Two-year MRI-defined structural damage and patient-reported outcomes following surgery or exercise for meniscal tears in young adults. Br J Sports Med. 2023 Nov 30;57(24):1566-1572. doi: 10.1136/bjsports-2023-107352. PMID 37879858
- [Derived] Damsted C, Thorlund JB, Holmich P, Lind M, Varnum C, Villumsen MD, Hansen MS, Skou ST. Effect of exercise therapy versus surgery on mechanical symptoms in young patients with a meniscal tear: a secondary analysis of the DREAM trial. Br J Sports Med. 2023 May;57(9):521-527. doi: 10.1136/bjsports-2022-106207. Epub 2023 Mar 6. PMID 36878666
- [Derived] Skou ST, Lind M, Holmich P, Jensen HP, Jensen C, Afzal M, Jorgensen U, Thorlund JB. Study protocol for a randomised controlled trial of meniscal surgery compared with exercise and patient education for treatment of meniscal tears in young adults. BMJ Open. 2017 Aug 21;7(8):e017436. doi: 10.1136/bmjopen-2017-017436. PMID 28827270